CLINICAL TRIAL: NCT02418299
Title: Prospective, Single Centre Study of Er:YAG Laser Treatment for Female Stress and Mixed Urinary Incontinence (IncontiLase)
Brief Title: Er:YAG Laser Treatment for Female Stress and Mixed Urinary Incontinence (IncontiLase)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Juna d.o.o. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J013
Record Dates: First submitted 2015-04-08; First posted 2015-04-16 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Female Stress Urinary Incontinence; Mixed Incontinence, Urge and Stress
Keywords: urinary incontinence; Er:YAG laser
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IncontiLase Er:YAG laser treatment (Experimental): Er:YAG laser treatment for stress and mixed urinary incontinence
  Interventions: Device: IncontiLase Er:YAG laser treatment

INTERVENTIONS:
Device: IncontiLase Er:YAG laser treatment — Each patient will receive 2-3 sessions of Er:YAG laser treatment for stress and mixed urinary incontinence (IncontiLase)
  Other Names: IncontiLase

SUMMARY:
The purpose of this study was to evaluate the effect of a non-invasive Er:YAG thermal laser therapy in treating female stress and mixed urinary incontinence.

DETAILED DESCRIPTION:
Urinary incontinence (UI) is a common disorder that affects women of various ages and impacts all aspects of life. Therapeutic approaches range from conservative therapy, which is heavily dependent on patient compliance, to different, more invasive, surgical procedures.

The aim of the study was to evaluate the non-invasive erbium:yttrium-aluminum-garnet (Er:YAG) laser treatment (IncontiLase) as a potential treatment strategy for stress UI (SUI) and mixed UI (MUI). The treatment works by thermally affecting vaginal mucosa, with an emphasis on the anterior vaginal wall, resulting with partial denaturation of collagen fibres and stimulation if new collagen formation, all of which leads to firmer support for the urethra and the improvement of incontinence symptoms.

The investigators included 175 women with newly diagnosed SUI (66% of women) and MUI (34 %), respectively and performed on average 2.5±0.5 procedures in each woman separated by a two-month period, using Er:YAG laser. Patients were clinically examined and classified by incontinence types (SUI and MUI) and grades (mild, moderate, severe and very severe) using International Consultation on Incontinence Modular Questionnaire (ICIQ) and assessing Incontinence Severity Index (ISI): ISI before the therapy was 5.7±2.1 points. Treatment discomfort was measured at every session with visual analogue system pain scale, and adverse effects and patients' satisfaction were followed. Follow-ups were performed at two, six and twelve months after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* clinically confirmed UI
* normal PAP smear (Papanicolaou cytology)
* negative urine culture
* integrity of the vaginal mucosa (without injuries or bleeding)

Exclusion Criteria:

* pregnancy
* intake of photosensitive drugs
* vaginal injuries or vaginal bleeding
* infection in the treated area
* clinical diagnosis of pure urge urinary incontinence

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2012-03; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change in the Incontinence Severity Index (ISI) calculated from the ICIQ-UI short form questionnaire | at baseline and 2, 6 and 12 months after treatment

SECONDARY OUTCOMES:
VAS index for the assessment of pain | at baat baseline and 2, 6 and 12 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Urška Bizjak-Ogrinc, Dr, Principal Investigator — Juna d.o.o.

REFERENCES:
- See also: The Juna Clinic — http://www.juna.si